CLINICAL TRIAL: NCT03566173
Title: Association Between Nonalcoholic Fatty Liver Disease and Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ningbo5
Record Dates: First submitted 2018-05-25; First posted 2018-06-25 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Acute Pancreatitis; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Pancreatitis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The early evaluation of AP severity are vital. Previous studies have shown non-alcoholic fatty liver disease (NAFLD) is associated with severity of acute pancreatitis (AP). This study is aimed to investigate the relationship between NAFLD and AP severity.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is a potentially lethal disease capable of wide clinical variation. Severe acute pancreatitis (SAP) is devastating, with a mortality rate ranging from 10% to as high as 85%. So it's important to identify severe patients which require aggressive early treatment and prolonged specialist care. There are a lot of multifactorial scorings and specific laboratory tests in predicting AP severity, such as Ranson's, Acute Physiology and Chronic Health Examination (APACHE)-II, serum Interleukin-6 (IL-6), and C-reactive protein (CRP) level. However, they have limitations in predicting outcomes of AP patients. The biochemical markers are not accurate enough. Ranson's scores were calculated after 48 hours of admission. Their practical utilization as predictors of severity is tough. Novel prognostic biomarker is needed to further develop for prognosis in AP patients.

Nonalcoholic fatty liver disease (NAFLD) refers to fat deposition and oxidative stress of free radicals in hepatocytes. NAFLD is the most common chronic liver disease worldwide. The prevalence averages 30% in developed countries, and estimated to be 10% in developing countries. Its presentation ranges from asymptomatic steatosis to fibrosis, and cirrhosis with 3-5%. It is evident clinically with increased risk of developing obesity, cardiovascular diseases (CVD), hyperlipidaemia, and type 2 diabetes mellitus (T2DM). Acting as an endocrine organ, the liver is the source of adipokines and inflammatory cytokines. Alterations in the production and secretion are increased in patients with NAFLD. It is strongly related to insulin resistance (IR) and metabolic disorders. Previous studies noted that NAFLD is closely related to severity of AP. CT scans are usually performed at admission to diagnose AP severity, which are also helpful to assess NAFLD. It could act as a valuable prognostic factor in AP patients and help to recognize potential severe patients.

However, no clear pathways could explain the association between NAFLD and AP at present. Besides, the data is scarce. More research will pay more attention to this topic. In this study, the investigators investigated the association between NAFLD and AP.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with AP
2. age >18 years

Exclusion Criteria:

1. an age of <18 years
2. without complete data and CT scans
3. previous splenectomy or hepatectomy
4. a past history of AP
5. an ambiguous pancreatic margin

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis criteria for AP was defined as the presence of at least 2 of the 3 following factors: (1) abdominal pain characteristic of AP; (2) serum amylase and/or lipase levels≥3 times the upper limit of the normal level, and (3) characteristic findings of AP on a CT scanning.
Sampling Method: Non-Probability Sample
Enrollment: 1662 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Comparisons of variables (age in years, BMI in kg/m2, pancreas attenuation in HU) on the basis of AP severity | the physical examination data in the year of 2017
  Comparisons of variables on the basis of AP severity by one-way analysis of variance (ANOVA)

SECONDARY OUTCOMES:
Association between NAFLD and severity outcomes in AP patients | the physical examination data in the year of 2017
  Association between liver/spleen attenuation (L/S) ratio in Hounsfield units (HU) and severity outcomes in AP patients by Cox regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lei Xu, Dr, Principal Investigator — Department of gastroenterology,Ningbo No.1 Hospital, Ningbo, China
Locations (1):
- Ningbo NO.1 hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No